CLINICAL TRIAL: NCT06721117
Title: Investigation of Grip Strength, Pain and Anxiety Levels in Dentists
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Research Assisstant, Hacettepe University
Other Study IDs: SUBU 2
Record Dates: First submitted 2024-11-30; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Grip; Muscle Disorder; Pain, Chronic; Anxiety
Keywords: pain; pain thereshold
MeSH Terms: conditions — Muscular Diseases; Chronic Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dentists: The participants of the study will consist of dentists working at Sakarya Oral and Dental Health Hospital. The aim is to include 50 dentists in the study. The individuals to be included in the study will be selected by random lottery.
  Inclusion criteria; To have graduated from the Faculty of Dentistry To have 1 year or more professional experience
  Exclusion criteria; To have received physical therapy from any region in the last 6 months or to be currently receiving physical therapy, To have a congenital musculoskeletal deformity, To have a neurological or rheumatic disease, To have undergone surgery due to a musculoskeletal disorder.
  Interventions: Other: Grip strength assessment; Other: Forearm muscle strength assessment; Other: Pain threshold assessment; Other: Anxiety level assessment

INTERVENTIONS:
Other: Grip strength assessment — Jamar hand dynamometer, recommended by the American Hand Therapists Association and accepted as the gold standard in many studies due to its high validity and reliability, will be used to measure hand grip strength. Pinchmeter (Baseline Mechanical Pinch Gauge) will be used to measure fine grip strength. Hand grip and finger grip strength measurements will be made in the recommended standard position of sitting, shoulder adduction and neutral rotation, elbow 90 degrees flexed, forearm in mid-rotation and supported, wrist in neutral. In the test procedure, 3 measurements will be taken for hand grip and finger grip strengths with one-minute intervals between each measurement and the averages will be recorded.
Other: Forearm muscle strength assessment — Wrist isometric muscle strength assessment will be performed with a handheld dynamometer (Lafayette Instrument Company, Lafayette, Indiana, USA). Patients will be placed in the supine, prone and sitting positions using the positions required for the fine muscle test method defined by Lovett and will be performed without compensatory movements. Wrist flexor and extensor muscles will be assessed. The values obtained with isometric contraction will be recorded in kg. Muscle strength measurements will be assessed bilaterally, in three repetitions for 5 seconds. The average value of the three repetition results will be recorded.
Other: Pain threshold assessment — Pain sensitivity to pressure will be assessed with a pain measuring device called an algometer. The Baseline Dolorimeter brand algometer will be used in the assessment. 3 measurements will be taken from the "midpoint of the upper trapezius muscle" and "C7" points between the lateral edge of the acromion and C7. The areas will be marked before the measurement. The algometer will be placed perpendicular to these points. The patients will be asked to report the moment they first felt the pain and 30 seconds of rest will be given between the measurements. The value on the display will be read and the pain threshold will be recorded in pounds (1kg=2.2 pounds).
Other: Anxiety level assessment — The anxiety level will be determined with the Beck Anxiety Inventory. The Beck Anxiety Inventory is a scale developed by Aaron T. Beck (1988). This scale consists of 21 questions. For each item, the patient is asked to report how he/she has felt during the past week.
  The items are scored as 0, 1, 2 or 3. The score range is between 0-63. For the total score, < 21 is considered mild, 22-35 is considered moderate, and > 36 is considered severe. The Turkish validity study of the Beck anxiety scale was conducted by Ulusoy et al (1996).

SUMMARY:
The aim of the study is to evaluate the relationship between professional experience and grip strength, pain threshold and anxiety level in dentists. As a result of the results obtained, we aim to contribute an original study to the literature and to increase awareness by informing the dentists participating in the study.

DETAILED DESCRIPTION:
Our hypotheses:

H1: Professional experience has an effect on hand grip strength in dentists. H2: Professional experience has an effect on finger grip strength in dentists. H2: Professional experience has an effect on pain in dentists. H3: Professional experience has an effect on anxiety level in dentists.

The unique value of our study is that it is the first study to examine the relationship between dentists' professional experience and grip strength, pain, and anxiety. When we look at the literature, we have not found any studies examining the effect of dentists' professional experience on grip strength and pain. In the study, grip strength, pain threshold, and forearm grip strength will be evaluated. Grip strength will be assessed with a Jamar hand dynamometer, pinch grip with a Baseline brand pinchmeter, pain threshold with a dolorometer, and forearm grip strength with a handheld dynamometer. Anxiety will be assessed with the Beck Anxiety Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Graduating from the Faculty of Dentistry
* Having 1 year or more professional experience

Exclusion criteria;

* Having received physical therapy from any area in the last 6 months or currently receiving physical therapy,
* Having a congenital musculoskeletal deformity,
* Having a neurological or rheumatic disease,
* Having undergone surgery due to a musculoskeletal disorder.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants of the study will consist of dentists working at Sakarya Oral and Dental Health Hospital. The aim is to include 50 dentists in the study. "Informed Voluntary Consent" will be obtained from dentists who volunteer to participate in the study. Each participant will be asked to fill out demographic information and data collection forms. Demographic information collection will consist of questions regarding age, gender, weight, height, body mass index, smoking, alcohol use, and chronic disease information.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Handgrip assessment | up to one week
  Grip strength will be determined by evaluating the gross grip and pinch grip. A pinchmeter (Baseline Mechanical Pinch Gauge) will be used to measure the fine grip strength. The measurement of hand grip and finger grip strength will be made in the recommended standard position of sitting, shoulder adduction and neutral rotation, elbow 90 degrees flexed, forearm in mid-rotation and supported, wrist in neutral. In the test procedure, 3 measurements will be taken for hand grip and finger grip strength with one minute intervals between each measurement and the averages will be recorded.

SECONDARY OUTCOMES:
Forehand muscle strength assessment | up to one week
  Wrist isometric muscle strength assessment will be performed with a handheld dynamometer (Lafayette Instrument Company, Lafayette, Indiana, USA). Patients will be positioned in the supine, prone and sitting positions, using the positions required for the fine muscle testing method described by Lovett, and will be performed before compensatory movements occur. Wrist flexor and extensor muscles will be assessed. The values obtained with isometric contraction will be recorded in pounds.
Pain thereshold assessment | up to one week
  Pain sensitivity to pressure will be assessed with a pain measuring device called an algometer. The Baseline Dolorimeter brand algometer will be used in the assessment. 3 measurements will be taken from the "midpoint of the upper trapezius muscle" and "C7" points between the lateral edge of the acromion and C7. The areas will be marked before the measurement. The algometer will be placed perpendicular to these points. The patients will be asked to report the moment they first feel pain and 30 seconds of rest will be given between measurements. The value on the display will be read and the pain threshold will be recorded in pounds (1kg=2.2 pounds).
Anxiety level assessment | up to one week
  The anxiety level will be determined with the Beck Anxiety Inventory. The Beck Anxiety Inventory is a scale developed by Aaron T. Beck (1988). This scale consists of 21 questions. For each item, the patient is asked to report how he/she has felt during the past week.
  The items are scored as 0, 1, 2 or 3. The score range is between 0-63. For the total score, < 21 is considered mild, 22-35 is considered moderate, and > 36 is considered severe. The Turkish validity study of the Beck anxiety scale was conducted by Ulusoy et al (1996).

REFERENCES:
- [Derived] Arslan SG, Yildiz A, Gultekinler BD. Relationship between hand grip and pinch strength, body composition, pain threshold, and anxiety in dentists. Ir J Med Sci. 2025 Jun;194(3):939-947. doi: 10.1007/s11845-025-03941-4. Epub 2025 Mar 28. PMID 40153116